CLINICAL TRIAL: NCT02282371
Title: A Phase Ib Study of Cetuximab + BYL719 + IMRT (Intensity-Modulated Radiation Therapy) in Stage III/IVB Head and Neck Squamous Cell Cancer (HNSCC)
Brief Title: Cetuximab + BYL719 + IMRT (Intensity-Modulated Radiation Therapy) in Stage III/IVB Head and Neck Squamous Cell Cancer (HNSCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-116
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: Cetuximab; BYL719; IMRT (Intensity-Modulated Radiation Therapy); 14-116
MeSH Terms: interventions — Cetuximab; Alpelisib; Radiotherapy, Intensity-Modulated

ARMS (1):
- Cetuximab + BYL719 + IMRT (Experimental): Cetuximab loading dose, 400 mg/m2 intravenously (IV). IMRT, 1 fraction/day, up to total of approximately 70 Gy, over approximately 33 treatment days Cetuximab 250 mg/m2 weekly IV X 7 weeks Daily BYL719, according to dose escalation scheme followup clinic visits every 3 months for 2 years,every 6 months for the next 3 years, and annually thereafter.
  Interventions: Drug: Cetuximab; Drug: BYL719; Radiation: IMRT (Intensity-Modulated Radiation Therapy)

INTERVENTIONS:
Drug: Cetuximab
Drug: BYL719
Radiation: IMRT (Intensity-Modulated Radiation Therapy)

SUMMARY:
This is a phase 1b study, which means that the purpose of the study is to establish the maximum dose of a pill drug called BYL719, when given with a standard treatment for patients with head and neck squamous cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally and/or regionally advanced (M0) head and neck squamous cell carcinoma (AJCC Stage III-IVB), cytologically or pathologically confirmed by Department of Pathology at MSKCC, for which curative-intent radiation therapy is planned.
* Age ≥ 18 years
* ECOG Performance Status ≤ 1
* Adequate organ function and laboratory parameters as defined by:

  * Absolute neutrophil count ≥ 1.0 x 109/L
  * Hemoglobin ≥ 9 g/dl
  * Platelets ≥ 100 x 109/L
  * AST/SGOT and ALT/SGPT ≤ 2.5X ULN (upper limit of normal)
  * bilirubin ≤ 1.5X ULN
  * creatinine ≤ 1.5X ULN
  * Fasting glucose < 140 mg/dL
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for males at least 4 months thereafter and for females at least 3 months thereafter.
* Negative serum pregnancy test (β-hCG) within 72 hours before starting study treatment for all women of childbearing potential.
* Able to understand and voluntarily sign the informed consent form, and able to comply with the study visit schedule and other protocol requirements.
* Low risk for tumor lysis syndrome (TLS)
* Sexually active males must use a condom during intercourse while taking the drugs and for 16 weeks after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
* Patient is able to swallow and retain oral medication

Exclusion Criteria:

* Any prior known radiation therapy in head and neck area
* Clinically significant cardiac disease or impaired cardiac function such as:

  * Congestive heart failure (CHF) requiring treatment (New York Heart Association ≥ grade 2), Left Ventricular Ejection Fraction (LVEF) ≤ 50% dose determined by multi-gated acquisition (MUGA) scan or echocardiogram, or uncontrolled arterial hypertension defined by blood pressure greater than 140/80 mmHg at rest (average of 3 consecutive readings)
  * History or current evidence of clinically significant cardiac arrhythmias, atrial fibrillation and/or conduction abnormality, (e.g. congenital long QT syndrome, high grade\complete AV blockage).
  * Acute coronary syndrome (including myocardial infarction, unstable angina, coronary artery bypass graft (CABG), for coronary angiography angioplasty and stenting), < 3 months prior to screening
  * QT interval adjusted according to Fredericia (QTcF) > 480 msec on screening EKG
* Patient with clinically manifest diabetes mellitus, or documented steroid induced diabetes mellitus
* Patient with history of another malignancy within 2 years prior to starting study treatment, except for cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient who has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient who has had systemic therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study entry
* Patient who has undergone major surgery ≤ 4 weeks prior to starting study treatment or who has not recovered from side effects of such procedure
* Any other condition that would, in the investigator's judgment. preclude patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g. infection/inflammation, intestinal obstruction, social/psychological complications
* Impaired GI function or GI disease that may significantly alter the absorption of oral BYL719 (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Patient who has participated in a prior therapeutic investigational drug study within 30 days prior to enrollment
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patient is currently receiving treatment with drugs known to be strong inhibitors or inducers of isoenzyme CYP3A. The patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the start of treatment. Switching to a different medication prior to the start of treatment is allowed; (Refer to Appendix 2).
* Known positive serology for human immunodeficiency virus (HIV), active hepatitis B, and/or active hepatitis C infection
* Patient has a known hypersensitivity to any of the excipients of BYL719
* Patient has a known hypersensitivity to cetuximab or any other monoclonal antibody
* Patient has a known history of non-compliance to medical regimen or inability to grant consent
* Pregnant nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL)
* Women Patient who does not apply highly effective contraception during the study and through the duration as defined below after the final dose of study treatment:

  a. Sexually active males should use a condom during intercourse while taking drug and for 16 weeks after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid b. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 16 weeks after the final dose of study treatment. Highly effective contraception is defined as either: i. Total abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception].

ii. Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). [For female study subjects, the vasectomized male partner should be the sole partner for that patient] iv. Use a combination of the following (both a+b):

1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
3. Note: Hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as BYL719 may decrease the effectiveness of hormonal contraceptives.

Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago.

* Patients with nasopharyngeal carcinoma are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-10-30 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
determine the phase II-recommended dose of BYL719 | 2 years
  Patients will be treated in cohorts of size three to six and the dosage will be escalated if the clinical toxicity is acceptable.

SECONDARY OUTCOMES:
Adverse events | 2 years
  Adverse events (AEs) will be assessed according to NCI common toxicity criteria (CTC) version 4. DLT is defined as any toxicity requiring radiotherapy treatment delay of ≥ 7 calendar days, or any ≥ Grade 3 toxicity (other than those excluded from the DLT definition, below). Patients who require dose reduction in BYL719 due to toxicity will be deemed to have experienced DLT.

CONTACTS AND LOCATIONS:
Overall Officials: David Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/